CLINICAL TRIAL: NCT02896218
Title: Therapeutic Monitoring of Vancomycin in Critical Ill Patients: a Registry
Acronym: VCMTDMinCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Qinggang GE, M.D. Chief physician, Peking University Third Hospital
Other Study IDs: CM-001
Record Dates: First submitted 2016-08-17; First posted 2016-09-12 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Critically Ill
Keywords: Vancomycin; Critically Ill; Pharmacist; Population Pharmacokinetic; Bayesian Methods
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pharmacist consulting group: When physicians make the decision that patients need to prescribe vancomycin or need dose adjustment, they will call for a pharmacist consultation. Pharmacists will provide the initial regimen based on PPK methods if applicable, otherwise give the suggestion of the initial dosage according to guidelines. Also, pharmacists will give suggestions on the time of sampling for serum concentration measurement. For dosage adjustment, pharmacists will be informed the results of serum vancomycin concentration, and then make a calculation using Bayesian estimation to determine whether there is a necessity to change the dosing regimen. Pharmacists will follow the patients until they discharge.
  Interventions: Other: Pharmacists consultation
- Usual care group: Empirical use of vancomycin without pharmacists consultation.

INTERVENTIONS:
Other: Pharmacists consultation — Pharmacists consultation of vancomycin individualized dosing strategy
  Groups: Pharmacist consulting group

SUMMARY:
Vancomycin is a glycopeptide antibiotic that is the first line antibiotics for the treatment of serious gram-positive infections involving methicillin-resistant Staphylococcus aureus (MRSA). Its therapeutic window is narrow, so there is a need to monitor serum vancomycin concentration in clinical practice, especially in the critically ill patients. So far, few studies have investigated the clinical outcomes of the dosage strategy that vancomycin dosage is administered and adjusted individually using PPK and Bayesian methods based on observed concentrations. The objective of this study is to investigate the effectiveness, safety and economics of the vancomycin individualized dosing service provided by pharmacists.

DETAILED DESCRIPTION:
Vancomycin is a glycopeptide antibiotic that is the first line antibiotics for the treatment of serious gram-positive infections involving methicillin-resistant Staphylococcus aureus (MRSA). Vancomycin use is associated with several adverse events, including nephrotoxicity and ototoxicity. Its therapeutic window is narrow, so there is a need to monitor serum vancomycin concentration in clinical practice, especially in the critically ill patients. Moreover, the Chinese vancomycin TDM guideline recommended that vancomycin dosage should be administered and adjusted individually based on population pharmacokinetic(PPK) and Bayesian methods. However, there is a gap between clinical practice and the guideline. So far, few studies have investigated the clinical outcomes of the dosage strategy that vancomycin dosage is administered and adjusted individually using PPK and Bayesian methods. Pharmacists could provide the vancomycin individualized dosing service by joining the ICU multidisciplinary team. The objective of this study is to investigate the effectiveness, safety and economics of the vancomycin individualized dosing service provided by pharmacists.

This is a single-center, ambispective cohort study. Patients from the retrospective and prospective cohort will be divided into 2 groups by exposure. The exposure is whether patients received pharmacists' consultation. Patients who meet the inclusion and exclusion criteria will be included in our registry. As a non-intervention study, these information as below will be collected: basic demographics, diagnosis, the initial dosage regimen and adjusted strategy of vancomycin, combined special treatment and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to intensive care unit(ICU), Peking University Third Hospital since JAN 2010.
* Receiving vancomycin therapy for 72 hours or more.
* Aged ≥ 18 years.

Exclusion Criteria:

* Administration of vancomycin in non-intravenous access.
* Life expectancy of less than 24 hours.
* Pregnancy women.
* Presence of immunodeficiency.
* Presence of hematological disorder.
* Written informed consent not obtained in the prospective cohort.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The prospective cohort: all patients in this cohort will receive pharmacist consultation when prescribed vancomycin.
  The retrospective cohort: patients in this cohort received usual care from JAN 2010 to MAR 2015; patients in this cohort received pharmacist consultation from APR 2016 to JUL 2016.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The rate of treatment failure | 2016-9 to 2018-1

SECONDARY OUTCOMES:
All cause mortality | 2016-9 to 2018-1
Mortality caused by infections | 2016-9 to 2018-1
Mortality caused by gram-positive infections | 2016-9 to 2018-1
Adverse events related to vancomycin | 2016-9 to 2018-1
Nephrotoxicity related to vancomycin | 2016-9 to 2018-1
  According to KDIGO, AKI is defined by any of the following:
  * Increase in serum creatinine by ≥0.3 mg/dL (≥26.5 micromol/L) within 48 hours; or
  * Increase in serum creatinine to ≥1.5 times baseline, which is known or presumed to have occurred within the prior seven days; or
  * Urine volume <0.5 mL/kg/h for six hours.
  All adverse events will be assessed and analyzed with WHO-UMC causality criteria by investigators. Adverse events related to vancomycin, especially nephrotoxicity, will be analyzed.
Cost-effectiveness of pharmacist intervention | 2016-9 to 2018-1
  The outcome is the incremental cost of preventing one treatment failure infection-related mortality or nephrotoxicity.
Duration of using ventilator | 2016-9 to 2018-1
Vancomycin dosage | -2016-9 to 201

CONTACTS AND LOCATIONS:
Overall Officials: Qinggang Ge, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rybak MJ, Lomaestro BM, Rotschafer JC, Moellering RC Jr, Craig WA, Billeter M, Dalovisio JR, Levine DP. Therapeutic monitoring of vancomycin in adults summary of consensus recommendations from the American Society of Health-System Pharmacists, the Infectious Diseases Society of America, and the Society of Infectious Diseases Pharmacists. Pharmacotherapy. 2009 Nov;29(11):1275-9. doi: 10.1592/phco.29.11.1275. PMID 19873687
- [Background] Ye ZK, Chen YL, Chen K, Zhang XL, Du GH, He B, Li DK, Liu YN, Yang KH, Zhang YY, Zhai SD; Guideline Steering Group, the Guideline Development Group and the Guideline Secretary Group. Therapeutic drug monitoring of vancomycin: a guideline of the Division of Therapeutic Drug Monitoring, Chinese Pharmacological Society. J Antimicrob Chemother. 2016 Nov;71(11):3020-3025. doi: 10.1093/jac/dkw254. Epub 2016 Jul 11. PMID 27494905
- [Background] Matsumoto K, Takesue Y, Ohmagari N, Mochizuki T, Mikamo H, Seki M, Takakura S, Tokimatsu I, Takahashi Y, Kasahara K, Okada K, Igarashi M, Kobayashi M, Hamada Y, Kimura M, Nishi Y, Tanigawara Y, Kimura T. Practice guidelines for therapeutic drug monitoring of vancomycin: a consensus review of the Japanese Society of Chemotherapy and the Japanese Society of Therapeutic Drug Monitoring. J Infect Chemother. 2013 Jun;19(3):365-80. doi: 10.1007/s10156-013-0599-4. Epub 2013 May 15. No abstract available. PMID 23673472
- [Background] Pea F, Bertolissi M, Di Silvestre A, Poz D, Giordano F, Furlanut M. TDM coupled with Bayesian forecasting should be considered an invaluable tool for optimizing vancomycin daily exposure in unstable critically ill patients. Int J Antimicrob Agents. 2002 Nov;20(5):326-32. doi: 10.1016/s0924-8579(02)00188-7. PMID 12431867
- [Background] Smith C, Burley C, Ireson M, Johnson T, Jordan D, Knight S, Mason T, Massey D, Moss J, Williams K. Clinical trials of antibacterial agents: a practical guide to design and analysis. Statisticians in the Pharmaceutical Industry Working Party. J Antimicrob Chemother. 1998 Apr;41(4):467-80. doi: 10.1093/jac/41.4.467. PMID 9598778